CLINICAL TRIAL: NCT02908165
Title: Randomized Phase II Trial of Chemoembolization and Sorafenib: Comparison Between Continuous and Sequential Treatment Regimens
Brief Title: Randomized Phase II Trial of Chemoembolization and Sorafenib
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A future study will be taking place using the same patient population.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1601017096
Record Dates: First submitted 2016-09-06; First posted 2016-09-20 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A- continuous schedule (Experimental): Subjects with HCC randomized to group A
  Interventions: Drug: conventional TACE in combination with sorafenib, administered on a continuous schedule
- Group B- sequential schedule (Active Comparator): Subjects with HCC randomized to group B
  Interventions: Drug: conventional TACE in combination with sorafenib, administered on a sequential schedule

INTERVENTIONS:
Drug: conventional TACE in combination with sorafenib, administered on a continuous schedule — Patients assigned to Group A will begin sorafenib on a continuous schedule starting at 400mg BID from Cycle 1 Day 1, one week prior to cTACE treatment on Cycle 1 Day 8. After week 6, cTACE will be provided on demand (as needed, up to 4 treatments total in the first 4 cycles) at week 2 in subsequent cycles, and sorafenib will continue to be administered. Patients will be allowed to undergo dose adjustments of sorafenib as long as it remains above the ¼ dose (400mg QOD).
  Arms: Group A- continuous schedule
Drug: conventional TACE in combination with sorafenib, administered on a sequential schedule — Patients assigned to Group B will undergo cTACE up to 4 treatments within the first 4 cycles as needed prior to starting sorafenib. After it is determined that no further TACE treatment is necessary (via imaging and clinical assessment on follow-up), administration of sorafenib will begin on Day 1 of the following cycle. Dosing will begin at 400mg BID and maintained continuously provided no unmanageable toxicities develop, with follow-up assessments performed on week 6 of every 1-2 cycles as needed. Patients in Group B will also be allowed to undergo dose adjustments of sorafenib as long as it remains above the ¼ dose (400mg QOD).
  Arms: Group B- sequential schedule

SUMMARY:
The study will be a single-center, randomized Phase II study of conventional TACE in combination with sorafenib, given either continuously or sequentially, in patients with unresectable HCC. The primary variables will be tumor response (by MR Imaging) and plasma VEGF levels, prior to and after cTACE.

DETAILED DESCRIPTION:
Transcatheter arterial chemoembolization (TACE) is the most widely performed procedure for patients with unresectable HCC. Although TACE can induce tumor necrosis, tumor recurrence and metastasis is not uncommon and likely due to stimulation of angiogenesis immediately after TACE. Plasma VEGF levels are significantly elevated following TACE procedures, usually peaking 24 to 48 hours after treatment.

Sorafenib, a multikinase inhibitor, has been shown to increase survival in patients with advanced HCC, presumably due to its predominant and strong antiangiogenic activities thereby preventing tumor growth. However, despite its targeted approach, sorafenib is not without toxicities; consequently most patients are unable to remain on full dose throughout the course of their treatment.

Because of sorafenib's antiangiogenic properties, it has been suggested that sorafenib could be used in combination with TACE to counteract the post-TACE angiogenic release and therefore prevent or minimize the risk of tumor recurrence. The possible synergy between TACE and sorafenib has been tested in numerous clinical studies. Although the safety profile has been clearly established, the efficacy of this combination therapy has yet to be demonstrated. Several combination methods have been tested, i.e., continuously where sorafenib is administered before the first TACE and then continuously throughout the planned TACE treatments, or sequentially where sorafenib is administered after the completion of TACE (usually 4 days after). Here, the investigators postulate that the sequence of the combination could have a significant impact on patient outcomes. Specifically, the investigators hypothesize that the continuous method is superior to that of the sequential protocol because the presence of sorafenib before the first TACE will preempt the peak of angiogenesis from TACE. To that end, the investigators propose to measure VEGF levels serially in order to detect differences between the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable hepatocellular carcinoma with liver-predominant disease, or patients with hepatocellular carcinoma who refuse surgery. No more than 30% of the cohort should have macrovascular invasion and/or asymptomatic extrahepatic disease. Multifocal HCC is acceptable, no diffuse HCC with greater than 70% tumor burden.
* Patient is at least 18 years of age.
* ECOG performance status of 0-1.
* Child-Pugh class of A or B (up to 7).
* Adequate end-organ function as manifested by:
* Absolute neutrophil count of ≥ 1500/mm3 and platelets ≥ 50,000/mm3
* Creatinine ≤ 2.0 mg/dL
* AST, ALT < 8X ULN
* Total bilirubin of ≤ 3 mg/dL
* Albumin > 2.0 g/dL
* INR < 2.0
* Leukocyte count > 3000 cells/mm3
* Patients who have been treated with previous hepatic surgery, radiofrequency ablation (RFA), percutaneous ethanol injection (PEI), or cryoablation are eligible if target lesion(s) have not been treated and local therapy is completed at least 6 weeks prior to entry.
* Patients with HBV are eligible if controlled with medication. Patients with HCV must have completed treatment with sustained viral response before being eligible for study.
* Patients with asymptomatic HIV infection are not eligible.
* Willingness of male and female subjects, who are not surgically sterile or post-menopausal, to use reliable methods of birth control for the duration of the study and for 30 days after the last dose of study medication.
* Patient must have signed informed consent prior to registration on study.
* Resolution of all acute toxic effects of any prior local treatment to CTC adverse event Grade 1 or 0.
* At least one tumor lesion can be accurately measured in at least one dimension according to RECIST (Appendix D). The lesion has not been previously treated with local therapy (such as surgery, radiation therapy, RFA, PEI, or cryoablation) unless it has shown progression in the interim.

Exclusion Criteria:

* Patients unable to swallow oral medications.
* Prior embolization, systemic, or radiation therapy for HCC (liver), or patients who have taken sorafenib for greater than 2 weeks. Patients randomized to the sequential arm who started taking sorafenib within 2 weeks of the planned TACE procedure will have to stop sorafenib for 2 weeks before undergoing TACE. This will prevent a possible confounding effect of sorafenib on patients randomized to the sequential arm.
* Tumor burden in the liver exceeding 70%.
* Complete occlusion of the main portal venous system. Partial or branch portal vein occlusion allowed if without reversal of flow.
* Ascites refractory to diuretic therapy (minimal or trace ascites on imaging is acceptable).
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis, and T1). Any cancer curatively treated more than 3 years prior to entry is permitted.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* History of bleeding within the past 4 weeks (unless deemed by PI as clinically insignificant, as for example, a brief episode of epistaxis).
* Any contraindication to doxorubicin or mitomycin-C administration.
* Evidence of severe or uncontrolled systemic diseases.
* Congestive cardiac failure greater than NYHA class 2 (Appendix E), myocardial infarction within 6 months, active coronary artery disease, cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, unstable angina, or laboratory or clinical finding that in the view of the principal investigator makes it undesirable for the patient to participate in the study.
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* History of stroke or transient ischemic attack within 6 months prior to study enrollment.
* Inadequately controlled hypertension (defined as systolic blood pressure of > 150/100 mmHg on antihypertensive medications). Patients with treated hypertension are eligible. Patients noted to be hypertensive in our clinic, but with documented normal blood pressure in the office of their referring physician, close follow-up with their referring providers, and a plan for coordination between the referring physician and our team for management of blood pressure while on therapy, are eligible.
* Significant vascular disease (e.g. aortic aneurysm, aortic dissection, peripheral vascular disease).
* History of organ allograft
* Presence of grade 2 or higher hepatic encephalopathy.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an additional experimental drug.
* Evidence of bleeding diathesis or coagulopathy or on warfarin. Note: if a patient has been on Coumadin for a period of 1 month and has been stable, they may be accepted into the protocol.
* Presence of clinically evident central nervous system or brain metastases.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study.
* Pregnant (positive pregnancy test) or lactating.
* Inability to comply with the study and/or follow-up procedures.
* Life expectancy of less than 12 weeks.
* Patients with concomitant HIV infection or AIDS-related serious acute or chronic illness.
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of study results.
* Active clinically serious infections (greater than Grade 2)
* Patients with obvious and/or symptomatic extrahepatic disease. Findings of uncertain significance, such as lung lesions less than 10 mm in diameter or enlarged periportal lymph nodes will not exclude patients.
* Any contraindication to an arterial procedure such as impaired clotting tests (platelet count < 50,000/mm3 or prothrombin activity < 50%).
* Any contraindication to sorafenib administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Tumor Response using Response Evaluation Criteria in Solid Tumors (RECIST) | 54 weeks
  RECIST criteria for tumor response:
  * Complete response - complete disappearance of all target lesions
  * Partial response - at least 30% decrease in the sum of the longest diameter (LD) of the target lesions, taking as a reference the baseline sum LD.
  * Stable disease - all other cases.
  * Progressive disease - at least a 20% increase in the sum of the LD of the target lesions, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Tumor Response using mREcist if applicable | 54 weeks
  mRECIST criteria for tumor response:
  * Complete response -disappearance of any intratumoral arterial enhancement in all target lesions.
  * Partial response - at least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions.
  * Stable disease - Any cases that do not qualify for either partial response or progressive disease.
  * Progressive disease - An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started.
EASL criteria for tumor response | 54 weeks
  * Complete response - Complete disappearance of all viable tumoral area and no new lesions. No new lesions may evolve during a 4 week period after initial documentation of response.
  * Partial response - Greater than 50% reduction in viable tumoral area of all measurable lesions via uptake of contrast.
  * Stable disease - All other cases.
  * Progressive disease - Greater than or equal to 25% increase in tumoral area of one or more measurable lesions or the appearance of new lesions.

SECONDARY OUTCOMES:
Laboratory Evaluations: Vascular endothelial growth factor (VEGF) Correlations | baseline and 54 Weeks
  Plasma VEGF levels will be compared between the two study arms. VEGF-A, as well as VEGF-R1 and R2 concentrations will be obtained.
  VEGF concentrations will also be correlated with tumor response of target lesions as determined by imaging assessments, and with overall survival.
Overall survival (OS) | 54 weeks
  Overall survival (OS) will be measured from the initiation of therapy until the date of death. OS will be assessed for patients treated with continuous sorafenib and cTACE and compared to those treated with sequential cTACE and sorafenib.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Geschwind, Principal Investigator — Professor of Radiology and Biomedical Imaging
Locations (1):
- Smilow Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No